CLINICAL TRIAL: NCT01321554
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial of Lenvatinib (E7080) in 131I-Refractory Differentiated Thyroid Cancer
Brief Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Trial of Lenvatinib (E7080) in 131I-Refractory Differentiated Thyroid Cancer (DTC)
Acronym: SELECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E7080-G000-303; 2010-023783-41 (EudraCT Number)
Record Dates: First submitted 2011-03-10; First posted 2011-03-23 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2020-03

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- Lenvatinib (Randomization Phase) (Experimental): Participants randomly assigned in a 2:1 ratio to receive blinded study drug (lenvatinib or matching placebo) until documentation of disease progression (confirmed by IIR), development of unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Lenvatinib
- Placebo (Randomization Phase) (Placebo Comparator): Participants randomly assigned in a 2:1 ratio to receive blinded study drug (lenvatinib or matching placebo) until documentation of disease progression (confirmed by IIR), development of unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Placebo
- Lenvatinib 24 mg (OOL Lenvatinib Treatment Period) (Experimental): Participants will receive lenvatinib 24 mg, orally once daily until documentation of disease progression (confirmed by investigator's assessment), development of unacceptable toxicity, or withdrawal of consent. Placebo treated participants in the Randomization Phase who have progressive disease confirmed by IIR could request to receive lenvatinib treatment in the OOL Treatment Period.
  Interventions: Drug: Lenvatinib
- Lenvatinib 20 mg (OOL Lenvatinib Treatment Period) (Experimental): Participants will receive lenvatinib 20 mg, orally once daily until documentation of disease progression (confirmed by investigator's assessment), development of unacceptable toxicity, or withdrawal of consent. Placebo treated participants in the Randomization Phase who have progressive disease confirmed by IIR could request to receive lenvatinib treatment in the OOL Treatment Period.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 24 mg (two 10-mg and one 4-mg lenvatinib matched capsules) taken orally once daily, continuously. Dose interruptions or reductions were allowed for subjects who experienced treatment-related toxicity.
  Other Names: Lenvatinib (Lenvima, E7080)
  Arms: Lenvatinib (Randomization Phase); Lenvatinib 24 mg (OOL Lenvatinib Treatment Period)
Drug: Placebo — Matching placebo (two 10-mg and one 4-mg lenvatinib matched capsules) taken orally once daily, continuously.
  Arms: Placebo (Randomization Phase)
Drug: Lenvatinib — Lenvatinib 20 mg (two 10-mg capsules) taken orally once daily, continuously. Dose interruptions or reductions were allowed for subjects who experienced treatment-related toxicity.
  The dose of lenvatinib during the OOL Lenvatinib Treatment Period was 24 mg once daily from 03 Oct 2011 until 15 Feb 2013. The dose was lowered at the request of the Data Monitoring Committee to 20 mg on 16 Feb 2013. Thus, more subjects were treated with 24 mg starting dose and the treatment duration was longer for these participants than those whose starting dose was 20 mg.
  Other Names: Lenvatinib (Lenvima, E7080)
  Arms: Lenvatinib 20 mg (OOL Lenvatinib Treatment Period)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase 3 study to compare the progression free survival, overall response rate (ORR) and safety of participants treated with lenvatinib 24 mg by continuous once daily oral dosing versus placebo. The study is conducted in 3 phases: a Prerandomization Phase (screening and baseline period), a Randomization Phase (double-blind treatment period), and an Extension Phase (Optional Open Label (OOL) Lenvatinib Treatment Period and a follow-up period).

DETAILED DESCRIPTION:
Randomization Phase: Participants will receive blinded study drug (lenvatinib/placebo) in 2:1 ratio until documentation of disease progression (confirmed by independent imaging review), development of unacceptable toxicity, or withdrawal of consent. After having completed the primary analysis, subjects treated with lenvatinib who have not experienced disease progression may request to continue open label lenvatinib at the same dose, according to the clinical judgment of the investigator. Participants who discontinue treatment for any reason other than disease progression will be followed in the Randomization Phase until disease progression or start of another anticancer treatment; these participants then enter the Extension Phase for survival follow-up. Extension Phase: Participants in the placebo arm who have disease progression confirmed by IIR could request to enter the OOL Lenvatinib Treatment Period and receive lenvatinib treatment. Participants will receive lenvatinib treatment until disease progression (investigator's assessment), development of intolerable toxicity, or withdrawal of consent. Participants who had disease progression during the Randomization Phase and did not enter the OOL Lenvatinib Treatment Period and all participants who discontinued lenvatinib treatment in the OOL Lenvatinib Treatment Period will enter the follow-up period. Participants will be followed for survival, and all anticancer treatments will be recorded until the time of death.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically confirmed diagnosis of one of the following DTC subtypes: Papillary thyroid cancer (PTC) or follicular thyroid cancer (FTC).
2. Measurable disease according to (RECIST 1.1) and confirmed by central radiographic review.
3. 131 I-refractory/resistant disease.
4. Evidence of disease progression within 12 months prior to signing informed consent (+1 month screening window).
5. Prior treatment with 0 or 1 vascular endothelial growth-factor (VEGF) or vascular endothelial growth-factor receptors (VEGFR) targeted therapy.
6. Adequate renal, liver, bone marrow, and blood coagulation function, as defined in the protocol.

Exclusion criteria:

1. Anaplastic or medullary carcinoma of the thyroid
2. 2 or more prior VEGF/ VEGFR-targeted therapies
3. Received any anticancer treatment within 21 days or any investigational agent within 30 days prior to the first dose of study drug.

Inclusion criteria for OOL Lenvatinib Treatment Period :

Participants were eligible for lenvatinib treatment in the OOL Lenvatinib Treatment Period if the met the following criteria:

1. Placebo-treated participants in the Randomization Phase who had progressive disease (PD) confirmed by IIR, and who requested treatment with lenvatinib.
2. Participants who continued to satisfy specified inclusion and exclusion criteria as presented in the study protocol.
3. Participants with maximum interval between the day of confirmation of PD by IIR and Cycle 1/Day 1 of the OOL Lenvatinib Treatment Period of less than or equal to 3 months.
4. No systemic anticancer treatment during the interval between the day of confirmation of PD by the IIR and Cycle 1/Day 1 of the OOL Lenvatinib Treatment Period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2011-03-17 (Actual); Primary Completion 2013-11-15 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (155):
- United States (38):
  - Facility 1, Little Rock, Arkansas
  - Facility 1, La Jolla, California
  - Facility 1, Los Gatos, California
  - Facility 1, Mission Viejo, California
  - Facility 1, Orange, California
  - Facility 2, Orange, California
  - Facility 1, Sacramento, California
  - Facility 1, Torrance, California
  - Facility 1, Aurora, Colorado
  - Facility 1, Washington D.C., District of Columbia
  - Facility 1, Orlando, Florida
  - Facility 1, Weston, Florida
  - Facility 1, Chicago, Illinois
  - Facility 2, Chicago, Illinois
  - Facility 1, Indianapolis, Indiana
  - Facility 1, Lexington, Kentucky
  - Facility 1, Baltimore, Maryland
  - Facility 1, Boston, Michigan
  - Facility 2, Boston, Michigan
  - Facility 1, Detroit, Michigan
  - Facility 1, Lansing, Michigan
  - Facility 1, Minneapolis, Minnesota
  - Facility 1, Columbia, Missouri
  - Facility 1, Omaha, Nebraska
  - Facility 1, Lebanon, New Hampshire
  - Facility 1, Morristown, New Jersey
  - Facility 1, Neptune City, New Jersey
  - Facility 1, New York, New York
  - Facility 2, New York, New York
  - Facility 1, The Bronx, New York
  - Facility 1, Columbus, Ohio
  - Facility 1, Portland, Oregon
  - Facility 1, Philadelphia, Pennsylvania
  - Facility 2, Philadelphia, Pennsylvania
  - Facility 1, Houston, Texas
  - Facility 1, Seattle, Washington
  - Facility 1, Morgantown, West Virginia
  - Facility 1, Milwaukee, Wisconsin
- Argentina (3):
  - Facility 1, Rosario
  - Facility 1, San Miguel de Tucumán
  - Facility 1, San Salvador de Jujuy
- Australia (5):
  - Facility 1, Saint Leonards, New South Wales
  - Facility 1, Herston, Queensland
  - Facility 1, Hobart, Tasmania
  - Facility 1, Melbourne, Victoria
  - Facility 1, Heidelberg
- Facility 1, Vienna, Austria
- Belgium (3):
  - Facility 1, Brussels
  - Facility 1, Edegem
  - Facility 1, Namur
- Brazil (7):
  - Facility 1, Brasília
  - Facility 1, Joinville
  - Facility 1, Novo Hamburgo
  - Facility 1, Rio de Janeiro
  - Facility 1, Salvador
  - Facility 1, São Paulo
  - Facility 2, São Paulo
- Canada (4):
  - Facility 1, London, Ontario
  - Facility 1, Toronto, Ontario
  - Facility 1, Montreal, Quebec
  - Facility 1, Québec
- Chile (5):
  - Facility 1, Santiago
  - Facility 2, Santiago
  - Facility 3, Santiago
  - Facility 1, Temuco
  - Facility 1, Viña del Mar
- Facility 1, Olomouc, Czechia
- Facility 1, Odense, Denmark
- France (14):
  - Facility 1, Angers
  - Facility 1, Bordeaux
  - Facility 1, Caen
  - Facility 1, Clermont-Ferrand
  - Facility 1, Dijon
  - Facility 1, Lille
  - Facility 1, Lyon
  - Facility 1, Marseille
  - Facility 1, Nice
  - Facility 1, Paris
  - Facility 2, Paris
  - Facility 1, Strasbourg
  - Facility 1, Vandœuvre-lès-Nancy
  - Facility 1, Villejuif
- Germany (7):
  - Facility 1, Essen
  - Facility 1, Hanover
  - Facility 1, Leipzig
  - Facility 1, Mainz
  - Facility 1, München
  - Facility 1, Tübingen
  - Facility 1, Würzburg
- Italy (16):
  - Facility 1, Catania
  - Facility 1, Livorno
  - Facility 1, Milan
  - Facility 2, Milan
  - Facility 3, Milan
  - Facility 4, Milan
  - Facility 5, Milan
  - Facility 1, Monserrato
  - Facility 1, Napoli
  - Facility 1, Padua
  - Facility 1, Pisa
  - Facility 1, Roma
  - Facility 2, Roma
  - Facility 1, Rozzano
  - Facility 1, Torino
  - Facility 1, Viagrande
- Japan (6):
  - Eisai Trial Site 1, Nagoya, Aichi-ken
  - Eisai Trial Site 2, Nagoya, Aichi-ken
  - Eisai Trial Site 1, Kashiwa, Chiba
  - Eisai Trial Site 1, Fukui-shi, Fukui
  - Eisai Trial Site 1, Kobe, Hyōgo
  - Eisai Trial Site 1, Koto-ku, Tokyo
- Poland (3):
  - Facility 1, Gliwice
  - Facility 1, Kielce
  - Facility 1, Poznan
- Portugal (2):
  - Facility 1, Lisbon
  - Facility 1, Porto
- Romania (3):
  - Facility 1, Bucharest
  - Facility 2, Bucharest
  - Facility 1, Cluj-Napoca
- Russia (4):
  - Facility 1, Krasnodar
  - Facility 1, Kursk
  - Facility 1, Obninsk
  - Facility 1, Ufa
- South Korea (6):
  - Facility 1, Daejeon
  - Facility 1, Gyeonggi-do
  - Facility 1, Seoul
  - Facility 2, Seoul
  - Facility 3, Seoul
  - Facility 1, Uijeongbu-si
- Spain (10):
  - Facility 2, Málaga, Andalusia
  - Facility 1, Barcelona, Catalonia
  - Facility 1, A Coruña, Galicia
  - Facility 2, Barcelona
  - Facility 1, L'Hospitalet de Llobregat
  - Facility 1, Madrid
  - Facility 2, Madrid
  - Facility 3, Madrid
  - Facility 4, Madrid
  - Facility 5, Madrid
- Sweden (3):
  - Facility 1, Gothenburg
  - Facility 1, Lund
  - Facility 1, Stockholm
- Thailand (5):
  - Facility 1, Bangkok
  - Facility 2, Bangkok
  - Facility 1, Chiang Mai
  - Facility 1, Khon Kaen
  - Facility 1, Pathumwan
- United Kingdom (8):
  - Facility 1, Aberdeen
  - Facility 1, Glasgow
  - Facility 2, London
  - Facility 3, London
  - Facility 1, Manchester
  - Facility 2, Manchester
  - Facility 1, Sheffield
  - Facility 1, Sutton

REFERENCES:
- [Derived] Taylor MH, Takahashi S, Capdevila J, Tahara M, Leboulleux S, Kiyota N, Dutcus CE, Xie R, Robinson B, Sherman S, Habra MA, Elisei R, Wirth LJ. Correlation of Performance Status and Neutrophil-Lymphocyte Ratio with Efficacy in Radioiodine-Refractory Differentiated Thyroid Cancer Treated with Lenvatinib. Thyroid. 2021 Aug;31(8):1226-1234. doi: 10.1089/thy.2020.0779. Epub 2021 Apr 29. PMID 33637020
- [Derived] Tahara M, Kiyota N, Hoff AO, Badiu C, Owonikoko TK, Dutcus CE, Suzuki T, Ren M, Wirth LJ. Impact of lung metastases on overall survival in the phase 3 SELECT study of lenvatinib in patients with radioiodine-refractory differentiated thyroid cancer. Eur J Cancer. 2021 Apr;147:51-57. doi: 10.1016/j.ejca.2020.12.032. Epub 2021 Feb 19. PMID 33611104
- [Derived] Tahara M, Brose MS, Wirth LJ, Suzuki T, Miyagishi H, Fujino K, Dutcus CE, Gianoukakis A. Impact of dose interruption on the efficacy of lenvatinib in a phase 3 study in patients with radioiodine-refractory differentiated thyroid cancer. Eur J Cancer. 2019 Jan;106:61-68. doi: 10.1016/j.ejca.2018.10.002. Epub 2018 Nov 22. PMID 30471649
- [Derived] Tahara M, Schlumberger M, Elisei R, Habra MA, Kiyota N, Paschke R, Dutcus CE, Hihara T, McGrath S, Matijevic M, Kadowaki T, Funahashi Y, Sherman SI. Exploratory analysis of biomarkers associated with clinical outcomes from the study of lenvatinib in differentiated cancer of the thyroid. Eur J Cancer. 2017 Apr;75:213-221. doi: 10.1016/j.ejca.2017.01.013. Epub 2017 Feb 24. PMID 28237867
- [Derived] Robinson B, Schlumberger M, Wirth LJ, Dutcus CE, Song J, Taylor MH, Kim SB, Krzyzanowska MK, Capdevila J, Sherman SI, Tahara M. Characterization of Tumor Size Changes Over Time From the Phase 3 Study of Lenvatinib in Thyroid Cancer. J Clin Endocrinol Metab. 2016 Nov;101(11):4103-4109. doi: 10.1210/jc.2015-3989. Epub 2016 Aug 22. PMID 27548104
- [Derived] Kiyota N, Schlumberger M, Muro K, Ando Y, Takahashi S, Kawai Y, Wirth L, Robinson B, Sherman S, Suzuki T, Fujino K, Gupta A, Hayato S, Tahara M. Subgroup analysis of Japanese patients in a phase 3 study of lenvatinib in radioiodine-refractory differentiated thyroid cancer. Cancer Sci. 2015 Dec;106(12):1714-21. doi: 10.1111/cas.12826. Epub 2015 Nov 2. PMID 26426092
- [Derived] Schlumberger M, Tahara M, Wirth LJ, Robinson B, Brose MS, Elisei R, Habra MA, Newbold K, Shah MH, Hoff AO, Gianoukakis AG, Kiyota N, Taylor MH, Kim SB, Krzyzanowska MK, Dutcus CE, de las Heras B, Zhu J, Sherman SI. Lenvatinib versus placebo in radioiodine-refractory thyroid cancer. N Engl J Med. 2015 Feb 12;372(7):621-30. doi: 10.1056/NEJMoa1406470. PMID 25671254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 117 investigative sites in Europe, North America, Asia Pacific, Japan, and Latin America from 17 March 2011 to 19 March 2019.
Pre-assignment Details: A total of 612 participants were screened for entry into the study. Of these 612 participants, 220 participants were screening failures and 392 participants were randomly assigned to receive either lenvatinib or placebo in a 2:1 ratio.
Groups:
- Randomization Phase: Lenvatinib 24 mg: Participants received lenvatinib 24 milligram (mg), hard capsule, orally, once daily, until documentation of disease progression (confirmed by Investigator-Initiated Research [IIR]), development of unacceptable toxicity, or withdrawal of consent.
- Randomization Phase: Placebo: Participants received matching-placebo, hard capsule, orally, once daily until documentation of disease progression (confirmed by IIR), development of unacceptable toxicity, or withdrawal of consent.
- OOL, Treatment Period: Lenvatinib 24 mg: Participants received lenvatinib 24 mg, hard capsule, orally, once daily in Treatment Period. Placebo treated participants in the Randomization Phase who had progressive disease confirmed by IIR, and who requested treatment with lenvatinib. OOL refers to Optional Open-Label.
- OOL, Treatment Period: Lenvatinib 20 mg: Participants received lenvatinib 20 mg, hard capsule, orally, once daily in Treatment Period. Placebo treated participants in the Randomization Phase who had progressive disease confirmed by IIR, and who requested treatment with lenvatinib.
Period: Randomization Phase
Arm/Group | Randomization Phase: Lenvatinib 24 mg | Randomization Phase: Placebo | OOL, Treatment Period: Lenvatinib 24 mg | OOL, Treatment Period: Lenvatinib 20 mg
Started | 261 | 131 | 0 | 0
Completed | 261 | 131 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: OOL Lenvatinib Treatment Period
Arm/Group | Randomization Phase: Lenvatinib 24 mg | Randomization Phase: Placebo | OOL, Treatment Period: Lenvatinib 24 mg | OOL, Treatment Period: Lenvatinib 20 mg
Started | 0 | 0 | 85 (Participants from randomization phase were re-randomized to OOL, treatment period.) | 30 (Participants from randomization phase were re-randomized to OOL, treatment period.)
Completed | 0 | 0 | 85 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomization Phase: Lenvatinib 24 mg: Participants received lenvatinib 24 mg, hard capsule, orally, once daily, until documentation of disease progression (confirmed by IIR), development of unacceptable toxicity, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Randomization Phase: Lenvatinib 24 mg | Randomization Phase: Placebo | Total
Number analyzed (Participants) | 261 | 131 | 392
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 62.1 (10.57) | 61.5 (10.09) | 61.9 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 56 | 192
  Male | 125 | 75 | 200

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of disease progression or death (whichever occurred first), as determined by blinded IIR using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 for the double-blind treatment period (Randomization Phase). Disease progression per RECIST v1.1 was defined as at least a 20 percent (%) relative increase and 5 millimeter (mm) absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study), recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: Date of randomization to the date of disease progression or death (whichever occurred first), assessed up to data cutoff date (15 Nov 2013) or up to approximately 2.5 years
Population: The full analysis set (Intent-to-Treat Analysis Set) included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: Lenvatinib 24 mg | Randomization Phase: Placebo
Number analyzed (Participants) | 261 | 131
months | 18.3 [15.1 to NA] — The upper limit of the 95% confidence interval was not estimable because an insufficient number of participants reached the event at the final assessment time point. | 3.6 [2.2 to 3.7]
Statistical Analysis 1: Comparison: Randomization Phase: Lenvatinib 24 mg vs Randomization Phase: Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 0.21, 99% CI 2-sided [0.14 to 0.31]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR, defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) as determined by blinded IIR using RECIST 1.1 for target lesions and assessed by magnetic resonance imaging/computed tomography (MRI/CT) scans (for double blind treatment period i.e. Randomization Phase). CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR = CR + PR.
Time Frame: as for outcome 1
Population: The full analysis set (Intent-to-Treat Analysis Set) included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomization Phase: Lenvatinib 24 mg | Randomization Phase: Placebo
Number analyzed (Participants) | 261 | 131
percentage of participants | 64.8 [59.0 to 70.5] | 1.5 [0.0 to 3.6]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival measured from the date of randomization until date of death from any cause. Overall survival is adjusted with rank preserving structural failure time.
Time Frame: Date of randomization until date of death from any cause, assessed up to data cutoff date (15 Nov 2013) or up to approximately 2.5 years
Population: The full analysis set (Intent-to-Treat Analysis Set) included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomization Phase: Lenvatinib 24 mg | Randomization Phase: Placebo
Number analyzed (Participants) | 261 | 131
months | NA [22.0 to NA] — The median OS was not yet reached for either the lenvatinib or the placebo arm (including crossover participants) at data cutoff date. | NA [14.3 to NA] — The median OS was not yet reached for either the lenvatinib or the placebo arm (including crossover participants) at data cutoff date.

4. Secondary Outcome: Pharmacokinetic (PK) Profile of Lenvatinib: Area Under the Plasma Concentration Curve
Time Frame: Cycle 1 Days 1 and 15: 0-10 hours postdose; Cycle 2 Day 1: 0-12 hour postdose
Population: The PK analysis set included all the participants who received at least one dose of study drug and had evaluable PK data.
Measure: Median (Full Range); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Randomization Phase: Lenvatinib 24 mg
Number analyzed (Participants) | 260
nanogram*hour per milliliter (ng*h/mL) | 3490 [1410 to 10700]

ADVERSE EVENTS:
Time Frame: For each participant, from the first dose till 30 days after the last dose up to approximately 8 years
Description: Safety was assessed by the monitoring and recording of all adverse events (AEs) and serious adverse events (SAEs); regular monitoring of hematology, clinical chemistry, and urine values; physical examinations; and regular measurement of vital signs, electrocardiograms (ECG), and echocardiograms.
Groups:
- OOL, Treatment Period: Lenvatinib 24 mg: Participants received lenvatinib 24 mg, hard capsule, orally, once daily in Treatment Period. Placebo treated participants in the Randomization Phase who had progressive disease confirmed by IIR, and who requested treatment with lenvatinib.
Arm/Group | Randomization Phase: Lenvatinib 24 mg | Randomization Phase: Placebo | OOL, Treatment Period: Lenvatinib 24 mg | OOL, Treatment Period: Lenvatinib 20 mg
All-Cause Mortality (participants affected / at risk) | 161/261 | 13/16 | 62/85 | 15/30
Serious Adverse Events (participants affected / at risk) | 171/261 | 31/131 | 62/85 | 16/30
Other Adverse Events (participants affected / at risk) | 259/261 | 118/131 | 84/85 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomization Phase: Lenvatinib 24 mg (N=261) | Randomization Phase: Placebo (N=131) | OOL, Treatment Period: Lenvatinib 24 mg (N=85) | OOL, Treatment Period: Lenvatinib 20 mg (N=30)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (5) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 5 (7) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aneurysm ruptured (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (4) | 0 (0) | 2 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (6) | 0 (0) | 3 (4) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 2 (3) | 1 (2) | 1 (1) | 0 (0)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Device failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 1 (3) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Gallbladder mucocoele (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 9 (9) | 0 (0) | 2 (3) | 1 (1)
Gallbladder perforation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device breakage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Diabetic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (12) | 5 (7) | 3 (5) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess soft tissue (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 7 (9) | 0 (0) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 6 (6) | 2 (3) | 1 (1) | 0 (0)
Testicular abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 10 (11) | 0 (0) | 1 (1) | 1 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (8) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 0 (0) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Laryngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lung infection (Infections and infestations) | 4 (6) | 0 (0) | 1 (3) | 2 (2)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (4) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (2) | 1 (2) | 0 (0)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Osmotic demyelination syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 12 (14) | 3 (3) | 5 (5) | 2 (3)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postictal paralysis (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 2 (3) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 2 (2) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
seizure (Nervous system disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Phlebitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic pulmonary embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomization Phase: Lenvatinib 24 mg (N=261) | Randomization Phase: Placebo (N=131) | OOL, Treatment Period: Lenvatinib 24 mg (N=85) | OOL, Treatment Period: Lenvatinib 20 mg (N=30)
Lymphopenia (Blood and lymphatic system disorders) | 20 (60) | 2 (2) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Platelet count decreased (Investigations) | 17 (108) | 0 (0) | 2 (2) | 5 (7)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (4)
Hypothyroidism (Endocrine disorders) | 14 (26) | 0 (0) | 7 (7) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 17 (30) | 2 (2) | 6 (7) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 18 (20) | 0 (0) | 5 (5) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 8 (12) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 31 (60) | 6 (13) | 7 (11) | 3 (11)
Oral pain (Gastrointestinal disorders) | 26 (44) | 1 (3) | 5 (9) | 0 (0)
Urinary tract infection (Infections and infestations) | 30 (54) | 7 (9) | 6 (8) | 3 (4)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Toothache (Gastrointestinal disorders) | 18 (22) | 5 (5) | 7 (8) | 2 (3)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 6 (7) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (22) | 6 (7) | 5 (5) | 1 (3)
Anxiety (Psychiatric disorders) | 15 (16) | 5 (6) | 5 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 21 (33) | 0 (0) | 8 (9) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 23 (33) | 15 (19) | 6 (8) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 27 (53) | 2 (3) | 9 (26) | 1 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 25 (83) | 3 (4) | 7 (84) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 38 (74) | 0 (0) | 11 (23) | 3 (6)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 6 (11) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 34 (39) | 7 (7) | 9 (14) | 6 (8)
Glossodynia (Gastrointestinal disorders) | 18 (32) | 0 (0) | 9 (12) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 (31) | 5 (5) | 11 (15) | 5 (13)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 32 (40) | 13 (14) | 11 (14) | 3 (5)
Pyrexia (General disorders) | 41 (58) | 15 (17) | 10 (20) | 5 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 43 (86) | 2 (2) | 9 (13) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47 (65) | 21 (29) | 16 (26) | 5 (5)
Abdominal pain upper (Gastrointestinal disorders) | 46 (85) | 11 (11) | 11 (13) | 9 (11)
Dry mouth (Gastrointestinal disorders) | 46 (58) | 11 (13) | 11 (12) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 12 (14) | 9 (10) | 3 (4)
Dysgeusia (Nervous system disorders) | 48 (70) | 4 (4) | 10 (13) | 6 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 51 (95) | 6 (9) | 12 (16) | 9 (16)
Dry skin (Skin and subcutaneous tissue disorders) | 32 (35) | 8 (8) | 10 (11) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 38 (66) | 6 (6) | 11 (14) | 3 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 27 (50) | 2 (2) | 12 (17) | 1 (3)
Dizziness (Nervous system disorders) | 45 (77) | 13 (14) | 15 (19) | 8 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 48 (73) | 9 (13) | 12 (27) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 36 (58) | 1 (1) | 14 (20) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 52 (81) | 12 (14) | 18 (29) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 55 (81) | 2 (4) | 14 (16) | 6 (8)
Oedema peripheral (General disorders) | 65 (124) | 10 (12) | 18 (20) | 3 (8)
Dysphagia (Gastrointestinal disorders) | 34 (47) | 9 (10) | 15 (15) | 3 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 46 (60) | 11 (13) | 14 (27) | 4 (6)
Abdominal pain (Gastrointestinal disorders) | 50 (109) | 5 (10) | 20 (34) | 8 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 85 (148) | 9 (15) | 19 (39) | 12 (25)
Headache (Nervous system disorders) | 105 (223) | 15 (21) | 19 (28) | 10 (35)
Cough (Respiratory, thoracic and mediastinal disorders) | 77 (114) | 24 (36) | 23 (30) | 8 (13)
Constipation (Gastrointestinal disorders) | 83 (113) | 20 (26) | 25 (32) | 5 (8)
Proteinuria (Renal and urinary disorders) | 99 (604) | 4 (5) | 26 (126) | 12 (24)
Asthenia (General disorders) | 69 (209) | 18 (29) | 21 (43) | 10 (26)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 86 (268) | 1 (1) | 24 (85) | 9 (44)
Stomatitis (Gastrointestinal disorders) | 100 (246) | 9 (10) | 28 (50) | 13 (22)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 87 (135) | 7 (8) | 33 (55) | 10 (13)
Vomiting (Gastrointestinal disorders) | 100 (217) | 19 (24) | 36 (67) | 9 (19)
Fatigue (General disorders) | 116 (298) | 33 (45) | 35 (64) | 13 (28)
Nausea (Gastrointestinal disorders) | 127 (295) | 34 (48) | 34 (67) | 12 (31)
Decreased appetite (Metabolism and nutrition disorders) | 148 (352) | 24 (31) | 43 (86) | 11 (24)
Weight decreased (Investigations) | 142 (450) | 20 (22) | 44 (101) | 18 (49)
Diarrhoea (Gastrointestinal disorders) | 182 (740) | 22 (27) | 55 (263) | 21 (66)
Hypertension (Vascular disorders) | 181 (720) | 19 (36) | 52 (84) | 21 (69)
Flatulence (Gastrointestinal disorders) | 15 (18) | 1 (1) | 3 (4) | 2 (6)
Malaise (General disorders) | 17 (29) | 0 (0) | 5 (8) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 18 (29) | 3 (3) | 5 (5) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 20 (23) | 3 (3) | 5 (8) | 0 (0)
Haematuria (Renal and urinary disorders) | 18 (22) | 3 (4) | 6 (9) | 0 (0)
Blood creatinine increased (Investigations) | 25 (54) | 2 (2) | 6 (8) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 24 (29) | 3 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 22 (31) | 3 (3) | 5 (7) | 3 (3)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 19 (36) | 2 (3) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 26 (40) | 7 (9) | 5 (10) | 3 (4)
Nasopharyngitis (Infections and infestations) | 28 (54) | 8 (8) | 6 (7) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 41 (78) | 5 (5) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 13 (23) | 8 (8) | 3 (3) | 2 (3)
Leukopenia (Blood and lymphatic system disorders) | 15 (47) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 20 (25) | 4 (4) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 14 (16) | 4 (5) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 17 (24) | 2 (2) | 5 (13) | 2 (3)
Influenza (Infections and infestations) | 16 (17) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 18 (31) | 1 (1) | 7 (9) | 2 (2)
White blood cell count decreased (Investigations) | 14 (47) | 4 (4) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 (28) | 2 (2) | 6 (13) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (25) | 3 (6) | 5 (11) | 1 (1)
Paraesthesia (Nervous system disorders) | 14 (18) | 4 (8) | 2 (2) | 3 (4)
Dysuria (Renal and urinary disorders) | 15 (17) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (25) | 6 (6) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 6 (11) | 3 (5)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 4 (7) | 2 (5)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 11 (13) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (5)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other